CLINICAL TRIAL: NCT05371730
Title: A Trial to Evaluate the Safety and Efficacy of NK Cells in Subjects With Myelodysplastic Syndromes
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nuwacell Biotechnologies Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Xiaoyu Zhu, M.D., Ph.D., Chief Physician, The First Affiliated Hospital of University of Science and Technology of China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AF/SC-12/02.0
Record Dates: First submitted 2022-05-07; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Relapsed / Refractory Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NK cells (Experimental)
  Interventions: Drug: NCR300

INTERVENTIONS:
Drug: NCR300 — Intravenous infusion of NK cells（NCR300）

SUMMARY:
A clinical study to Evaluate the Safety and Efficacy of NK cells in the treatment of Myelodysplastic Syndromes

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center pilot study. In this study, 15 patients will be enrolled. The primary purpose is to explore the safety including incidence of adverse events and serious adverse events.The secondary purpose is to explore the efficacy.

ELIGIBILITY:
Key Inclusion Criteria

1. Subjects should voluntarily participate in this clinical study, are fully aware of the study, have signed the Informed Consent Forms, and are willing to follow and able to complete all trial procedures.
2. Subjects who are more than 18 years old (including 18 years old), and less than 75 years old (including 75 years old).
3. Subjects who are diagnosed as Myelodysplastic Syndromes(MDS) according to the IWG 2016 diagnosis criteria.
4. Subjects who are diagnosed as relapsed or refractory MDS according to the IWG 2006 response criteria.
5. Subjects who don't accept nor be suitable for HSCT.
6. With the expected survival phase>3 months, subjects whose performance status scores of the Eastern Cooperative Oncology Organization (ECOG) are≤3.
7. Except for the exclusion of blood transfusion and granulocyte-stimulating factor drugs, the subjects should meet the following conditions :Hemoglobin（HGB）> 60g/L,platelet count（PLT）> 30 × 10^9 / L, white blood cell count（WBC）> 1.0 × 10^9 / L,neutrophil（ NE）> 0.5 × 10^9 / L.

"8.Organ function should meet the following criteria: Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and total bilirubin(TBIL) ≤ 2 times the upper limit of normal (ULN)； serum creatinine（Scr）≤ 1.5 times ULNl ;international normalized ratio(INR)≤ 2 times ULNl or activeated partial thromboplasting time(APTT)≤ 1.5 times ULNl ." 9.According to the Common Terminology Criteria for Adverse Event ( CTCAE ) Version 4.0 ,all of AEs caused by pre-treatment have returned to the grade 1.

Key Exclusion Criteria

1. Bone marrow blasts>20%.
2. Bone marrow fibrosis in diagnostic bone marrow biopsy.
3. Subjects who have received immunosuppressive therapy (such as antithymocyte globulin,Cyclosporine,Mycophenolate mofetil ,Sirolimus,Etanercept,Alemtuzumab etc.) or thrombopoietin receptor agonists (such as Romiplostim,Herombopag Olamine,Recombinant Human TPO etc.) within 1 month before enrollment.
4. Subjects who have received HSCT or other organ transplantations.
5. Subjects who have uncontrolled active systemic fungal, bacterial or viral infections.
6. When the virological test during the screening period shows that any of the following is met:positive test for the human immunodeficiency virus antibody, Hepatitis B surface antigen (HBsAg) and / or Hepatitis B core antibody (anti-HBc) and hepatitis B virus deoxyribonucleic acid > 10^3 copies / mL, Hepatitis C antibody (anti-HCV) or Treponema pallidum specific antibody(TPHA).
7. Subjects who are known to be allergic to the study drug and/or main components and/or any excipients of the study drug.

"8.Serious organ dysfunction or disease involving the heart, kidney, or liver, such as Respiratory failure.

New York Heart Association classification stage II, III, or IV congestive heart failure,QT interval prolongation,decompensated liver or renal insufficiency,uncontrolled hypertension ( > 160 / 100mmHg ) and dyslipidemia despite active treatment." 9.Active thrombosis,subjects who have a history of cardiovascular or cerebrovascular thrombotic events within 12 months.

10.Subjects who have had other uncured tumors within 5 years. 11.Subjects who have participated in any other clinical trials within 1 month before screening (excluding those who failed the screening or did not use study drugs for other reasons).

12.Subjects who have a history of alcohol, drug use or drug abuse. 13.Subjects who have a history of mental disorder. 14.Subjects who have potential health or social status (such as other severe, acute, chronic diseases laboratory abnormalities etc.) that may increase the risk of participating in the study and receiving the study drug, or may interfere with the interpretation of study results.

15.Pregnant women, lactating women, women of childbearing age who do not take appropriate contraceptive measures during the trial period (sterilization, intrauterine device, oral contraceptives or barrier contraception).

16.Subjects who are judged by the investigator to be unsuitable to participate in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
AE or SAE | From infusion day 365
  The incidence of AE or SAE of NK cells infusion

SECONDARY OUTCOMES:
Bone Marrow Morphology | 58 days after initial infusion
  The proportion of bone marrow blasts after NK cells infusions.
Objective response rate (ORR) | 58 days after initial infusion
  ORR (sum of CR and PR) after NK cells infusions